CLINICAL TRIAL: NCT07385989
Title: A Randomized Controlled Multicenter Phase 2 Clinical Trial of Golidocitinib Combined With P-GemOx Plus PD-1 Inhibitor Versus P-GemOx Plus PD-1 Inhibitor in the Treatment of First-Line Newly Diagnosed Advanced Extranodal NK/T-Cell Lymphoma (ENKTL) or Non-Nasal Extranodal NK/T-Cell Lymphoma (ENKTL)
Brief Title: Golidocitinib Combined With P-GemOx Plus PD-1 Inhibitor Versus P-GemOx Plus PD-1 Inhibitor in First-Line Newly Diagnosed Advanced or Non-Nasal Extranodal NK/T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: WEI XU (Other)
Responsible Party: Sponsor-Investigator, WEI XU, Chief Physician, Department of Hematology, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-682
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golidocitinib + P-GemOx + PD-1 Inhibitor (Experimental): Golidocitinib (150 mg orally once daily, Days 1-21) Pegaspargase (2000 U/m² intravenously, Day 2) Gemcitabine (1000 mg/m² intravenously, Day 1) Oxaliplatin (100 mg/m² intravenously, Day 1) PD-1 inhibitor (200 mg intravenously, Day 1) Participants receive 6 cycles of induction therapy; those achieving complete response (CR) or partial response (PR) will continue maintenance therapy (Golidocitinib + PD-1 inhibitor, same dosage/schedule) for 1 year or until disease progression.
  Interventions: Drug: Golidocitinib in combination with P-GEMOX and PD-1 inhibitor
- P-GemOx + PD-1 Inhibitor (Active Comparator): Pegaspargase (2000 U/m² intravenously, Day 2) Gemcitabine (1000 mg/m² intravenously, Day 1) Oxaliplatin (100 mg/m² intravenously, Day 1) PD-1 inhibitor (200 mg intravenously, Day 1) Participants receive 6 cycles of induction therapy; those achieving complete response (CR) or partial response (PR) will continue maintenance therapy (PD-1 inhibitor alone, same dosage/schedule) for 1 year or until disease progression.
  Interventions: Drug: PD-1 inhibitor in combination with P-GEMOX

INTERVENTIONS:
Drug: Golidocitinib in combination with P-GEMOX and PD-1 inhibitor — Participants receive this combination for 6 cycles of induction therapy. Those achieving complete response (CR) or partial response (PR) post-induction will continue maintenance therapy with golidocitinib plus PD-1 inhibitor (same dosage and administration schedule) for 1 year, or until disease progression, unacceptable toxicity, or voluntary withdrawal from the study. This regimen is designed to target the STAT3 signaling pathway (via golidocitinib) while combining cytotoxic chemotherapy (P-GEMOX) and immune checkpoint inhibition (PD-1 inhibitor) for synergistic anti-lymphoma activity.
  Arms: Golidocitinib + P-GemOx + PD-1 Inhibitor
Drug: PD-1 inhibitor in combination with P-GEMOX — Participants receive this combined regimen for 6 cycles of induction therapy. For those achieving complete response (CR) or partial response (PR) post-induction, maintenance therapy is continued with PD-1 inhibitor alone (same 200 mg intravenous dose on Day 1 of each 21-day cycle) for 1 year, or until disease progression, unacceptable treatment-related toxicity, or study discontinuation. This regimen represents a currently established first-line therapeutic option for advanced/non-nasal ENKTL, serving as the active comparator for evaluating the added benefit of golidocitinib in the experimental arm.
  Arms: P-GemOx + PD-1 Inhibitor

SUMMARY:
This is a multicenter, randomized, Phase 2 clinical trial designed to evaluate the efficacy and safety of golidocitinib combined with the P-GemOx (pegaspargase + gemcitabine + oxaliplatin) regimen plus PD-1 inhibitor, compared with P-GemOx plus PD-1 inhibitor alone, in participants with first-line newly diagnosed advanced (Stage III-IV) or non-nasal extranodal natural killer/T-cell lymphoma (ENKTL). Eligible participants will be randomly assigned 1:1 to two groups:

Experimental group: Golidocitinib (150 mg orally once daily, Days 1-21 per 21-day cycle) + P-GemOx (pegaspargase 2000 U/m² on Day 2; gemcitabine 1000 mg/m² on Day 1; oxaliplatin 100 mg/m² on Day 1, per 21-day cycle) + PD-1 inhibitor (200 mg intravenously on Day 1 per 21-day cycle).

Control group: P-GemOx + PD-1 inhibitor (same dosage/schedule as the experimental group, without golidocitinib). All participants will receive 6 cycles of induction therapy. Those achieving CR or partial response (PR) after induction will receive maintenance therapy for 1 year: the experimental group will continue golidocitinib + PD-1 inhibitor, while the control group will receive PD-1 inhibitor alone (both per 21-day cycles). The primary outcome is the complete response rate (CRR) after 6 induction cycles (assessed per the 2014 Lugano Classification for Lymphoma). Secondary outcomes include overall response rate (ORR), 2-year progression-free survival (PFS), 2-year overall survival (OS), and the incidence of treatment-related adverse events (graded per NCI-CTCAE Version 5.0). 40 participants will be enrolled across multiple Chinese medical centers. This Phase 2 trial will provide preliminary evidence to determine whether the golidocitinib combination regimen is a safe and effective first-line option for advanced or non-nasal ENKTL.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provides written informed consent (ICF) prior to any study procedures.
2. Aged 18-70 years (inclusive), regardless of sex.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histologically confirmed extranodal NK/T-cell lymphoma (ENKTL), staged as Stage III-IV or non-nasal ENKTL (per 2016 WHO Classification of Hematopoietic and Lymphoid Tumors).
5. At least one measurable/evaluable lesion (per 2014 Lugano Classification: measurable lesion ≥1.5 cm in longest diameter + ≥1.0 cm in shortest diameter; evaluable lesion with FDG uptake higher than liver on PET/CT).
6. Treatment-naive (no prior anti-cancer therapy for ENKTL).
7. Adequate organ function:

   AST/ALT ≤2.5×upper limit of normal (ULN); Total bilirubin (TBIL) ≤1.5×ULN; Serum creatinine <1.5×ULN or creatinine clearance (CrCl, via Cockcroft-Gault formula) ≥60 mL/min.
8. Reproductive-aged females have a negative pregnancy test at screening; all participants use effective contraception during the study and for 12 months after the last dose.
9. Expected survival ≥6 months.

Exclusion Criteria:

1. Complicated by hemophagocytic lymphohistiocytosis (HLH) or aggressive NK-cell leukemia.
2. Contraindication to golidocitinib, PD-1 inhibitor, or any component of the P-GEMOX regimen.
3. Lymphoma involvement of the central nervous system (CNS).
4. Major surgery (excluding diagnostic biopsy) within 4 weeks prior to study treatment initiation.
5. History of other malignant tumors (except curatively treated in situ cancers, e.g., cervical carcinoma in situ) within 5 years.
6. Uncontrolled severe comorbidities (e.g., NYHA Class II+ heart failure, unstable angina, myocardial infarction within 1 year, uncontrolled arrhythmias).
7. Active bleeding (e.g., gastrointestinal hemorrhage, cerebral hemorrhage).
8. Uncontrolled infection (requiring parenteral anti-infective therapy) within 7 days prior to study treatment.
9. Active hepatitis B/C: HBsAg+/HBcAb+ with HBV-DNA >2500 copies/mL (or 500 IU/mL); HCV antibody+ with positive HCV-RNA.
10. HIV infection or acquired immunodeficiency syndrome (AIDS).
11. Conditions impairing drug absorption (e.g., inability to swallow tablets, malabsorption syndrome).
12. Pregnant/lactating females, or reproductive-aged participants refusing contraception.
13. Psychiatric illness precluding informed consent or study compliance.
14. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) After 6 Cycles of Induction Therapy | Within 21 days after the completion of the 6th cycle of induction therapy (Each cycle is 21 days)
  The proportion of evaluable participants who achieve complete response (CR) following 6 cycles of induction therapy. CR is defined in accordance with the 2014 Lugano Classification for Lymphoma: this requires the complete disappearance of all measurable/evaluable lymphoma lesions, resolution of all disease-related clinical symptoms, and normalization of imaging findings (e.g., no residual measurable disease on CT/MRI, and no metabolically active disease on FDG-PET/CT). The analysis population is restricted to participants who complete at least 4 cycles of induction therapy and have available post-treatment efficacy assessment data.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) After 6 Cycles of Induction Therapy | Within 21 days after the completion of the 6th cycle of induction therapy At the end of Cycle 1 (each cycle is 28 days)
  The proportion of evaluable participants who achieve objective response (defined as complete response [CR] or partial response [PR]) following 6 cycles of induction therapy. Response assessment adheres to the 2014 Lugano Classification for Lymphoma: PR requires a ≥50% reduction in the sum of the longest diameters of measurable lesions, with no new lesions or progression of existing non-measurable disease. The analysis population includes participants who complete at least 4 induction cycles and have available post-treatment efficacy evaluation data.
2-Year Progression-Free Survival (PFS) | Up to 2 years after randomization
  The duration from randomization to the first occurrence of disease progression (per the 2014 Lugano Classification) or death from any cause. PFS will be estimated using the Kaplan-Meier method, and between-arm comparisons will be conducted via the log-rank test. Participants without progression or death at the end of follow-up will be censored at their last documented disease-evaluation date.
2-Year Overall Survival (OS) | Up to 2 years after randomization
  The duration from randomization to death from any cause. OS will be estimated using the Kaplan-Meier method, with between-arm comparisons performed using the log-rank test. Participants who remain alive at the 2-year follow-up endpoint will be censored at their last confirmed survival date.
Incidence of Treatment-Related Adverse Events (TRAE) | From the first dose of study intervention to 30 days after the last dose of study intervention
  The proportion of participants experiencing any treatment-related adverse event, graded per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. This includes the incidence of grade 3-4 TRAEs and serious adverse events (SAEs; defined as events that are life-threatening, require hospitalization, result in persistent disability, or are fatal).

IPD SHARING:
Plan to Share IPD: Undecided